CLINICAL TRIAL: NCT06996275
Title: Attachment and Post-traumatic Stress Disorder in Military Personnel: Characterisation of the French Military Population, Exploration of Biopsychosocial Factors and Study of the Impact of Reassuring Primers on Emotional Contagion Skills.
Brief Title: Attachment and Post-Traumatic Stress Disorder in Military Personnel: Characterization of the French Military Population, Exploration of Biopsychosocial Factors, and Study of the Impact of Security Priming on Emotional Contagion Capacities
Acronym: AT-HOME
Status: Not yet recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2024PBMD03; 2025-A00068-41 (Other: ID-RCB)
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Post-traumatic Stress Disorder (PTSD); Emotional Contagion
Keywords: PTSD; complex PTSD; military veteran; emotional contagion; oxytocin; vasopressine
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Salivary samplings : (i) for the measurement of vasopressin and oxytocin levels , via saliva impregnation by leaving an absorbent (cylindrical cotton) in the mouth for 2 minutes without chewing, and (ii) and for the analysis of genetic polymorphisms, by collecting 2 ml of spit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PTSD-group: military personnel or veterans suffering from PTSD
- no PTSD-group: military on active duty without PTSD

SUMMARY:
Post-traumatic stress disorder (PTSD) is a pathology that impairs the quality of life of sufferers. In military personnel, it can lead to military incapacity. This psychopathology is characterized by confrontation with one or more traumatic events in the individual's life history. Symptoms include cognitive and mood disorders, avoidance, hyperactivation (hypervigilance and anger) and intrusions (flashbacks and nightmares).

Studies show that the prevalence of PTSD in military personnel fluctuates considerably from one situation to another (pre-deployment/post-deployment, etc.). In these at-risk populations, the often more complex PTSD clinic may also account for the heterogeneity of prevalences observed. Nevertheless, PTSD tends to become chronic in military personnel, making it particularly difficult to return to a "previous" state. In French casualties, beyond the symptoms already mentioned, complaints focus on difficulties in social interaction situations involving others in social life (attachment style to others) and in everyday life (public transport, supermarket shopping, social interactions, presence of crowds...).

In the context of post-traumatic stress disorder, we would like to explore the processes of social cognition that enable people to interact in their environment, in relation to biological, psychosocial and physiological variables that may constitute risk or maintenance factors for the pathology.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria Common to Both Groups:

* Volunteers who agreed to participate in the study and provided written consent
* Affiliated with social security
* Proficient in the French language

Inclusion Criteria Specific to the "Military Personnel with PTSD" Group:

* Military personnel diagnosed with post-traumatic stress disorder related to their duties
* Participants in activities offered by the wounded service support units

Exclusion Criteria:

* Adults subject to a protective measure
* Refusal to participate in the study
* Unrectified Legionnaires

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: No-PTSD Group: Military personnel without PTSD will be recruited from within an infantry regiment of the army.
  PTSD Group: Military personnel with PTSD will be recruited during workshops conducted by the CABAT (Cellule d'Aide aux Blessés de l'Armée de Terre - Army Wounded Support Unit) in 2025 and 2026.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2025-05-27 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To characterize attachment styles within a military population by comparing a group of military personnel without PTSD (No-PTSD Group) with a group of military personnel with PTSD (PTSD Group). | One visit study
  Our primary outcome measure involves a comparison of the proportions of individuals exhibiting a secure attachment style versus an insecure attachment style (including the subtypes anxious-avoidant, anxious-ambivalent, and disorganized) between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Anaïs Duffaud, PhD, Study Director — Institut de Recherche Biomédicale des Armées

IPD SHARING:
Plan to Share IPD: No